CLINICAL TRIAL: NCT05694351
Title: GO EASY: Eating Habits and Physical Activity in Synergy for Diabetes Prevention in Families
Brief Title: Family-based Prevention of Diabetes Through Eating Habits and Physical Activity
Acronym: GO_EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Responsible Party: Principal Investigator, Svetlana Solgaard Nielsen, Principal Investigator, Occupational Therapist, PhD, postdoc, Slagelse Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 96452
Record Dates: First submitted 2022-12-29; First posted 2023-01-23 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Family Health; Health Behavior; Healthy Lifestyle; Prediabetic State; Telemedicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Behavior; Prediabetic State | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Families with type 2 diabetes (Experimental): Families (n=25) of at least two family members - minimum one adult and one child per family unit (appx. 100 individuals in total) will be included. A convenient study sample will be composed with no restriction to family types - traditional nuclear families, same-sex parenting families, single-parent families, or blended/ step-parent families). Balanced representation of different geographical areas within Region Zealand will be attempted.
  Interventions: Behavioral: Healthy meals and physical activity in families with type 2 diabetes

INTERVENTIONS:
Behavioral: Healthy meals and physical activity in families with type 2 diabetes — Families will participate in telehealth family education on diabetes management and prevention through lifestyle modifications in their everyday occupations regarding current recommendations for physical activity, grocery shopping, meal preparation, and family meal routines. Each family will be assisted in setting tailored goals for the family as a whole and individually regarding physical activity and dieting habits. The goals will be incorporated into family daily routines, to secure manageability and sustainability of the new lifestyle habits. Local facilities and communy networks will be engaged in this process to empower and motivate the participants. Working with the goals will be monitored and facilitated throughout the intervention period of 3 months. Before discharge, each family will co-produce a maintenance plan for physical activity and healthy dieting.
  Other Names: GO EASY: God ernæring og aktivitet for nye synergier i familier i Region Sjælland

SUMMARY:
Introduction: Type 2 diabetes represents a growing health risk for the society. An easy-access and low-cost intervention for the whole family will be developed to help families with (at risk of) type 2 diabetes maintain diabetes-frendly everyday life. The intervention will be tested for feasibility.

Methods: Following the framework for developing and conduct of complex interventions, the intervention will be developed on the basis of current evidence on family-based diabetes treatment and opinions of families with type 2 diabetes. The feasibility test will have embedded mixed methods one-group study design.

Participants: Families will answer a brief screening questionnaire. Families (n=25) that consist of at least one adult with (in risk of) type 2 diabetes living in the same household with at least one 5-18 yeard old child, and at least one family member living sedentary lifestyle, will participate.

Intervention: The 3-months long hybrid telehealth/face-to-face intervention with weekly 1-hour contacts with health professionals will deliver diabetes education and tailored support to implement more physical activity and healthy meals in the family everyday life. A 3-months long supervised maintenance phase with monthly professional contacts will be included.

Outcomes: Feasibility evaluation will be conducted using quantitative (quantifiable) and qualitative research methods. The feasibility data will be the primary outcomes of the study, collected and evaluated using the predefined research progression criteria applied the green-amber-red method. Sociodemography and secondary outcomes, such as physical activity, dieting habits, daily occupations, occupational balance, health and quality of life will be assessed at baseline and 3 and 6-months follow-ups. The quantitative results will be comprehended through qualitative data from participant interviews which will nuance the feasibility evaluation.

Analysis: Relevant statistical methods and qualitative analysis method will be applied.

Expected results: The intervention will help families achieve sustainable lifestyle changes, e.g., diabetes stabilized blood glucose in adults with type 2 diabetes, increased physical activity time and improved dieting habits, for better family health and well-being.

Ethics and dissemination: The trial does not have any obvious health risks for the participants. All the results - significant, non-significant and/ or inconclusive - will be reported.

DETAILED DESCRIPTION:
Note: T2D means type 2 diabetes

Design

The GO EASY intervention is an easy-access and low-cost intervention promoting physical activity and healthier meals in families with (at risk of) T2D. The intervention will be developed and tested for feasibility, following the recommendations on developing and conducting complex interventions from the Medical Research Council (MRC) framework.

Feasibility evaluation of the intervention will be conducted using quantitative (quantifiable) and qualitative research methods. The quantitative results will be comprehended through qualitative data which will help a nuanced in-depth evaluation of feasibility from participant and clinical perspectives.

For the quantitative (quantifiable) data collection on feasibility, predefined research progression criteria will be determined, and the green-amber-red method will be applied. The green-amber-red method with the categories GREEN (Proceed with the RCT/ implementation), AMBER (Proceed, but changes to the protocol need to be discussed and solved) and RED (Do not proceed unless the problem can be solved) will help evaluate the readiness of the intervention to be tested for effectiveness in an RCT. Parameters relevant to T2D research, i.e., dieting habits, routines, and physical activity, will be monitored and assessed before and after the intervention. Several families will participate in objective physical activity assessments using technological devices (activity trackers).

Min. 10 - max. 20 qualitative family interviews will study the mechanisms of what is at stake during changing health behavior within participating families. Families who earned the experiences with the activity tracker technology will be invited to share their experiences in a separate qualitative interview-based study in a walk-and-talk format to explore the acceptability and usability of the devices.

Data privacy and ethical concerns

The project follows the principles of The World Medical Association (WMA) described in the WMA Declaration of Helsinki. The ethical approval of the project is sought at The Regional Committee on Health Research Ethics in Region Zealand (Denmark). The Data Protection Agency in Region Zealand (reg.) and the Research & Innovation Organization (RIO) at the University of Southern Denmark (SDU) are sought for approval of the project. The use of activity trackers (Garmin) has been approved by the IT-Concern in Region Zealand.

The project procedures will be conducted in compliance with the European Union's (EU) General Data Protection Regulation (GDPR) and the Danish Data Protection Act. The project data may be used in other statistical and scientific projects approved by the internal (regional) data protection authorities or the Danish Data Protection Agency, with written permission from the main investigator for the current project. Other projects must report on data transmission from this project in their protocols. The transmitted data must be protected for identification of the individuals behind, e.g. by dissemination of the results. After project completion, all transmitted data must be archived and included in data collection in the definitive trial.

Biobank

A project biobank will be established in the Region Zealand Biobank for research purposes. Blood samples from adults with (at risk of) T2D will be obtained for monitoring blood glucose (Hb1Ac) before and after the intervention. The outcome is recommended for T2D studies and allows objective evaluation of health promotion planned in the research project. The biobank data is included in the applications sent to the Regional Committee on Health Research Ethics in Region Zealand, the Data Protection Agency in Region Zealand and the RIO at SDU.

Each blood sample will be attached to the personal project ID. Key codes will only be available for the research responsible during the ongoing research. By the end of the research activities (see the project timeline), all the biological materials used in the project and key codes will be destroyed. Subsequently, all the data will be anonymized and archived in Region Zealand. Anonymized excessive biological materials collected in this project will be stored in the Region Zealand Biobank for further unspecific research.

The participants will be informed of the blood sampling purpose and asked for their consent on delivering biological material to the biobank (see the project information leaflet and the informed consent form for adults). The consent will imply that relevant information from Hb1Ac analysis (values beyond the recommended range) will be registered in patient journal in Sundhedsplatformen with a note to the participant and his or her family physician right after obtaining the analysis results. Because monitoring of Hb1Ac is essential for T2D prevention, the participants will not be given the option to decline to receive the reports.

Risks and discomfort

The trial does not have any obvious health risks for the participants. Educated health professional assessors will supervise all the participants during assessment procedures.

Study setting

The Department for Physiotherapy and Occupational Therapy at Næstved-Slagelse-Ringsted Hospitals is leading and delivering the intervention in cooperation with SDCS. The six SDCS departments located in Slagelse, Næstved, and Holbæk will accommodate the intervention delivery.

Participants

Families (n=25) of at least two family members - minimum one adult and one child per family unit (appx. 100 individuals in total) will be included. A convenient study sample will be composed with no restriction to family types - traditional nuclear families, same-sex parenting families, single-parent families, or blended/ step-parent families). Balanced representation of different geographical areas within Region Zealand will be attempted.

Recruitment

The participants will be enrolled with help from already established research collaborators at the Department for Physiotherapy and Occupational Therapy at Næstved-Slagelse-Ringsted Hospitals who have contact to target population in general practice and municipal healthcare centers. Additionally, outpatient healthcare services for children and youth, local and social media, and public schools, will be involved.

Leaflets distributed through the study settings and news and social media will provide parents with contact information and access to a detailed project description and an invitation to an online information meeting in a secure VDX-video communication system, an educated project assistant will provide detailed oral information on participation. Phone or e-mail contacts will be answered by the project assistant. At least one week of thinking time will be given.

Families that have received detailed written and oral information on the project will be provided with access to a brief digital questionnaire designed for eligibility screening in the secure system RedCap. The eligibility screening shall be completed by each adult family member individually. The eligibility screening questionnaire will start with informed consent on participation in the project, before asking any questions on eligibility. Opened questionnaires with no consent will remain anonymous and registered as incomplete. Inconsistencies in the completed eligibility screening responses will be clarified by phone.

The informed consent will give the principal investigator and his representative access to information relevant to the project from journal records, e.g., medication lists, other treatments and adverse events, to ensure eligibility and support compliance during the intervention.

All the included families will participate in the intervention. Due to the study design and the intervention character, the participants, intervention deliverers, outcome assessors and statisticians cannot be blinded to treatment. A minimum of six participating families will be invited to the qualitative interviews after discharge from the intervention. Recruitment to the qualitative part of the study will be completed when data saturation is observed, expectedly at the maximum of ten family interviews.

Statistical considerations for the feasibility study

No sample size calculation will be performed. According to the rationale about feasibility, we considered a convenient sample of 25 families (appx. 100 individuals) would be sufficient to reach the boundaries in predefined research criteria and evaluate the intervention feasibility. Acceptable dropout of max. 20% is included in the sample size determined for this study. All the families will be invited to participate in the family interviews post-discharge. A minimum of 6 families will be attempted to be included in the family interviews to ensure data saturation.

Analysis

Quantitative analyses: According to the normality check results, the data will be described by mean ± SD or median (range) and analyzed for pre-post changes. Parametric or nonparametric statistics will be applied to the data analysis performed using the STATA 17.0 software (StataCorp, Texas, USA).

Qualitative analysis: The interview data will be transcribed verbatim and analyzed using thematic content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parents (aged 18 or older) with (or at risk of) type 2 diabetes living in the same household with 5-17 years old children
* At least one family member not meeting the current physical activity recommendations.

Exclusion Criteria:

* Pregnancy or postpartum period (6 months after birth)
* Current critical illness, e.g. cancer
* Participating in other type 2 diabetes treatment programs

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of the participants recruited per months | 3 months
  cf. predefined research progression criteria
Rate of the participants recruited per months | 6 months
  cf. predefined research progression criteria
Percentage of participants completed the intervention | 3 months
  cf. predefined research progression criteria
Percentage of participants completed the intervention | 6 months
  cf. predefined research progression criteria
Rate of participants' adherence to the intervention's sessions (attendance registration forms) | 3 months
  cf. predefined research progression criteria
Rate of participants' adherence to the intervention's sessions (attendance registration forms) | 6 months
  cf. predefined research progression criteria
Participants' self-perceived relevance (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  cf. predefined research progression criteria
Participants' self-perceived relevance (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  cf. predefined research progression criteria
Participants' self-perceived timing (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  cf. predefined research progression criteria
Participants' self-perceived timing (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  cf. predefined research progression criteria
Participants' self-perceived mode of delivery (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  cf. predefined research progression criteria
Participants' self-perceived mode of delivery (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  cf. predefined research progression criteria
Satisfaction with the treatment (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  cf. predefined research progression criteria
Satisfaction with the treatment (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  cf. predefined research progression criteria
Assessment procedure acceptance (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  cf. predefined research progression criteria
Assessment procedure acceptance (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  cf. predefined research progression criteria
Adverse events | 3 months
  cf. predefined research progression criteria
Adverse events | 6 months
  cf. predefined research progression criteria
Fidelity of delivery (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  cf. predefined research progression criteria
Fidelity of delivery (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  cf. predefined research progression criteria
Contextual appropriateness (questionnaire, 5-items Likert scale, higher score is best) | 3 months
  Treatment acceptance, cf. predefined research progression criteria
Contextual appropriateness (questionnaire, 5-items Likert scale, higher score is best) | 6 months
  Treatment acceptance, cf. predefined research progression criteria

SECONDARY OUTCOMES:
Weekly physical activity, self-reported | Change from baseline to 6 months
  physical activity time (hours and minutes)
Daily wake-time physical activity, objective | Change from baseline to 6 months
  Physical activity time (hours and minutes) using Axivity AX3 accelerometer mounted on the right thigh for 7 days
Daily walking steps, objective | Change from baseline to 6 months
  Step count using Axivity AX3 accelerometer mounted on the right thigh for 7 days
Dieting habits | Change from baseline to 6 months
  generic questionnaire, weekly consumption of greens, fruits, meat and fish, and alcohol
Glucaemic control | Change from baseline to 6 months
  Haemoglobin A1c blood test
BMI | Change from baseline to 6 months
  calculated by division of self-reported data on body weight in kilograms by height in meters squared (only adults)
Activities of daily living | Change from baseline to 6 months
  generic questionnaire, occupational performance problems (5-items Likert scale, higher score is worst)
Occupational balance | Change from baseline to 6 months
  OBQ13 questionnaire -13 items measured, 6-step ordinal scales (higher score is best)
Self-perceived health today | Change from baseline to 6 months
  EQ-5D-5L, EQ-VAS (0-100)
Health-related quality of life | Change from baseline to 6 months
  EQ-5D-5L, EQ-Index - 5 dimensions: (1) mobility; (2) self-care; (3) usual activities; (4) pain/discomfort and (5) anxiety/depression, & 5-level rating - Level 1: no problems; Level 2: slight problems; Level 3: moderate problems; Level 4: severe problems; Level 5: extreme problems (higher is worst)
Well-being | Change from baseline to 6 months
  WHO5 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Solgaard Nielsen, PhD, Principal Investigator — Slagelse Hospital
Locations (1):
- Svetlana Solgaard Nielsen, Slagelse, Denmark

IPD SHARING:
Plan to Share IPD: No